CLINICAL TRIAL: NCT04681066
Title: A Randomized, Double-Blind, Placebo Controlled Dose-Ranging Study of Auxora in Patients With Acute Pancreatitis and Accompanying Systemic Inflammatory Response Syndrome
Brief Title: A Study of Auxora in Patients With Acute Pancreatitis and Accompanying SIRS
Acronym: CARPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM4620-203
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Pancreatitis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Pancreatitis; Systemic Inflammatory Response Syndrome | interventions — zegocractin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2.0 mg/kg (1.25 mL/kg) (Active Comparator): administered intravenously over 4 hours at a constant rate of infusion. They will be administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Interventions: Drug: CM-4620 Injectable Emulsion or CM-4620-IE
- 1.0 mg/kg (0.625 mL/kg) (Active Comparator): administered intravenously over 4 hours at a constant rate of infusion. They will be administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Interventions: Drug: CM-4620 Injectable Emulsion or CM-4620-IE
- 0.5 mg/kg (0.3125 mL/kg) (Active Comparator): administered intravenously over 4 hours at a constant rate of infusion. They will be administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Interventions: Drug: CM-4620 Injectable Emulsion or CM-4620-IE
- Placebo (1.25, 0.625, or 0.3125 mL/kg) (Placebo Comparator): patients randomized to placebo will receive one of three following volumes (1.25 mL/kg, 0.625 mL/kg, and 0.3125 mL/kg. although three volumes - all patients randomized to placebo will be analyzed together as one arm. administered intravenously over 4 hours at a constant rate of infusion. They will be administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CM-4620 Injectable Emulsion or CM-4620-IE — Auxora is to be administered as an IV infusion and is supplied as a translucent, white to yellowish colored, sterile, non-pyrogenic emulsion containing 1.6 mg/mL of the active pharmaceutical ingredient CM4620. CM4620-IE is supplied as an 80 mL fill in a 100 mL, single-use glass vial. The drug product is formulated as an emulsion due to the low solubility of CM4620 in aqueous solution. CM4620-IE contains egg phospholipids, medium chain triglycerides, glycerin, edetate disodium salt dehydrate (EDTA), sodium hydroxide (as needed to adjust pH), and sterile water for injection.
  Other Names: Auxora
  Arms: 0.5 mg/kg (0.3125 mL/kg); 1.0 mg/kg (0.625 mL/kg); 2.0 mg/kg (1.25 mL/kg)
Other: Placebo — Matching Placebo is to be administered as an IV infusion and is supplied as a translucent, white to yellowish, sterile, non-pyrogenic emulsion carrier containing no active pharmaceutical ingredient. Placebo is supplied as an 80 mL fill in a 100 mL single-use vial. Placebo contains the same ingredients as Auxora except that it does not contain CM4620.
  Arms: Placebo (1.25, 0.625, or 0.3125 mL/kg)

SUMMARY:
Approximately 216 patients with acute pancreatitis and accompanying SIRS will be randomized at approximately 30 sites. Patients will be randomly assigned to either Auxora at one of three dose levels or one of three placebo volumes to maintain the double-blind. Study drug infusions will occur every 24 hours for three consecutive days for a total of three infusions. Patients will remain hospitalized as per standard of care and once discharged will be asked to complete a daily meal diary and return for a Day 30 safety assessment. It is recommended that patients randomized in the study should not be discharged from the hospital until solid food is tolerated, abdominal pain has resolved or been adequately controlled, and there is no clinical evidence of infection necessitating continued hospitalization.

DETAILED DESCRIPTION:
This double blind, randomized, placebo-controlled study will evaluate the efficacy, safety, and tolerability of three different dose levels of Auxora in patients with acute pancreatitis and accompanying SIRS.

Approximately 216 patients will be randomized 1:1:1:1 into one of 4 groups using a computer generated randomization scheme accessed through an interactive voice/web response system (IXRS). Randomization will be first stratified by gender (male or female) and then by risk for organ failure in the gender subgroups (higher or lower). Higher risk for organ failure is defined by the presence of both an elevated hematocrit (HCT ≥44% for men or ≥40% for women) and hypoxemia (imputed PaO2/FiO2 ≤360). Lower risk for organ failure is defined by the absence of either or both an elevated hematocrit and hypoxemia. The PaO2/FiO2 will be determined using an arterial blood gas or imputed using pulse oximetry.

All patients will have received a Screening CECT of the abdomen/pancreas before being randomized into the study. CECTs performed as standard of care may be used as the Screening CECT but must have been performed in the 24 hours before Consent or after Consent and before Randomization.

The Start of First Infusion of Study Drug (SFISD) should occur within 8 hours of the patient or LAR providing informed consent. Patients randomized to Group 1 will receive 2.0 mg/kg of Auxora intravenously every 24 hours (±1 hour) for a total of three doses. Patients randomized to Group 2 will receive 1.0 mg/kg of Auxora intravenously every 24 hours (±1 hour) for a total of three doses. Patients randomized to Group 3 will receive 0.5 mg/kg of Auxora intravenously every 24 hours (±1 hour) for a total of three doses. Patients randomized to Group 4 will receive emulsion without any active pharmaceutical ingredient. Patients in Group 4 will receive one of three randomly assigned dose volumes, 1.25 mL/kg, 0.625 mL/kg, or 0.3125 mL/kg, which will be administered intravenously every 24 hours (±1 hour) for a total of three doses. The dosing will be based on actual body weight obtained at the time of hospitalization or screening for the study. As described in the pharmacy manual, the upper limit of the volume of Auxora and volume of Placebo that will be administered will be 156.25 mL. The sponsor, investigators and patients will be blinded to the assigned group. In the event of a medical emergency, investigators will be able to receive the treatment assignment if required to provide optimal care of the patient.

For all 4 groups, a study physician or appropriately trained delegate will perform assessments at screening, at the baseline assessment, immediately prior to the SFISD, and then every 24 hours until 240 hours after the SFISD, or until discharge if earlier. If patients remain hospitalized at Day 12, assessments will then be performed every 48 hours starting on Day 12 until Day 28, or until discharge if earlier. Patients discharged from the hospital before Day 25 will return at Day 30 (+5 days) to perform the Day 30 assessments. If patients are discharged on Days 25-29, the Day 30 assessments may be performed prior to discharge.

Patients will receive another CECT of the abdomen/pancreas at the Day 30 (±5 days) visit. All CECTs performed as standard of care after randomization and before the Day 30 CECT will also be captured. A blinded central reader will read the Screening, Day 30, and any standard of care CECTs obtained between randomization and the Day 30 visit.

Patients will complete the modified American Neurogastroenterology and Motility Society Gastrointestinal Cardinal Symptom Index Daily Diary (mGCSI-DD) worksheet at the baseline assessment, at 96 hours, 168hours, Day 14 and Day 21 (for patients who remain hospitalized on these days), on the day of discharge, and daily at bedtime after discharge until the Day 30 visit. Patients who are discharged on Days 25-29 will not complete the mGCSI worksheet after discharge.

It is recommended that all patients randomized in the study should receive care consistent with the 2018 American Gastroenterological Association (AGA) Institute Technical Review of the Initial Medical Management of Acute Pancreatitis. Patients should receive local standard of care (SOC) for the management of other medical conditions.

In patients with acute pancreatitis, the AGA strongly recommends early oral feeding (within 24 hours) rather than keeping the patient nil per mouth (Nil per Os, NPO). Patients randomized into the study, therefore, will be offered a low fat, ≥500-calorie solid meal at each mealtime after the infusion of the first dose of study drug if alert and not on mechanical ventilation, or if not NPO for a planned surgery/medical procedure, or if not NPO because of an acute medical condition. If the patient does not wish to eat the solid meal when offered or is unable to tolerate the solid meal, they should then be offered a liquid meal. The same approach should occur at each subsequent mealtime. When patients eat a solid meal, it should be recorded if they ate ≥50% of the meal and if they either vomited or experienced an increase in abdominal pain in the two hours after eating a meal.

It is also recommended that all patients randomized in the study should not be discharged from the hospital until solid food is tolerated, abdominal pain has resolved or been adequately controlled, and there is no clinical evidence of infection. Tolerating solid food is defined as eating ≥50% of a low fat, ≥500-calorie solid meal without an increase in abdominal pain or vomiting. If the patient is not tolerating either solid or liquid meals, tube feedings should be considered.

All protocol required laboratory testing, except biomarker and PK samples, will be performed at the local laboratory. Results from the biomarkers and PK blood samples collected as part of the protocol and being tested at a central lab will not be available to assist the PI or treating physician in managing the patient.

ELIGIBILITY:
Inclusion Criteria:

All of the following must be met for a patient to be randomized into the study:

1. The diagnosis of acute pancreatitis has been established by the presence of abdominal pain consistent with acute pancreatitis together with at least 1 of the following 2 criteria:

   1. Serum lipase > 3 times the upper limit of normal (ULN);
   2. Characteristic findings of acute pancreatitis on abdominal imaging;
2. The diagnosis of SIRS has been established by the presence of at least two of the following four criteria:

   1. Temperature < 36°C or > 38°C;
   2. Heart rate > 90 beats/minute;
   3. Respiratory rate >20 breaths/minute or arterial carbon dioxide tension (PaCO2) <32 mmHg;
   4. White blood cell count (WBC) >12,000 mm3, or <4,000 mm3, or > 10% immature (band) forms;
3. At least one of the following criteria is also present:

   1. A peripancreatic fluid collection or a pleural effusion on a contrast-enhanced computed tomography (CECT) performed in the 24 hours before Consent or after Consent and before Randomization;
   2. Abdominal examination documenting either abdominal guarding or rebound tenderness;
   3. Hematocrit ≥44% for men or ≥40% for women;
4. The patient is ≥ 18 years of age;
5. Lack of pancreatic necrosis, pancreatic calcifications, pancreatic pseudocysts and no evidence for previous necrosectomy or pancreatic surgery identified by CECT performed in the 24 hours before Consent or after Consent and before Randomization;
6. A female patient of childbearing potential who is sexually active with a male partner is willing to practice acceptable methods of birth control for 180 days after the last dose of study drug. A female patient must not attempt to become pregnant for 180 days;
7. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 180 days after the last dose of study drug. A male patient must not donate sperm for 180 days;
8. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

Patients with any of the following conditions or characteristics must be excluded from randomizing:

1. Expected survival <6 months;
2. Suspected presence of cholangitis in the judgment of the treating physician;
3. The patient has a known history of:

   1. Organ or hematologic transplant;
   2. HIV, hepatitis B, or hepatitis C infection;
   3. Chronic pancreatitis;
4. Current treatment with:

   1. Chemotherapy;
   2. Immunosuppressive medications or immunotherapy
   3. Pancreatic enzyme replacement therapy;
   4. Hemodialysis or Peritoneal Dialysis;
5. The patient is known to be pregnant or is nursing;
6. The patient has participated in another study of an investigational drug or therapeutic medical device in the 30 days before randomization;
7. Allergy to eggs or known hypersensitivity to any components of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-reported gender
Enrollment: 216 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Study Director — CalciMedica, Inc.
Locations (37):
- United States (27):
  - Long Beach Medical Center, Long Beach, California
  - LA County Hospital - USC, Los Angeles, California
  - Cedars Sinai, Los Angeles, California
  - University of California at Irvine Medical Center, Orange, California
  - Harbor UCLA Medical Center, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - The Stamford Hospital, Stamford, Connecticut
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Northwestern University Hospital, Chicago, Illinois
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Missouri School of Medicine, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northshore University Hospital, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - Regional One Health, Memphis, Tennessee
  - John Peter Smith Hospital, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Health Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - CAMC Institute for Academic Medicine, Charleston, West Virginia
- India (10):
  - SPMC, Bīkaner
  - PGIMER, Chandigarh, Chandigarh
  - Malla Reddy Narayana, Hyderabad
  - MDM Hospital, Jodhpur
  - Lisie Hospital, Kochi
  - Seven Star Hospital, Nagpur
  - JIPMER, Puducherry
  - MTES' Sanjeevan Hospital, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - IGMU (India Gandhi Medical), Shimla

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Auxora 2.0 mg/kg (1.25 mL/kg): High dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
  CM-4620 Injectable Emulsion (CM4620-IE): Auxora is administered as an IV infusion and is supplied as a sterile, non-pyrogenic emulsion containing 1.6 mg/mL of the active pharmaceutical ingredient CM4620. CM4620-IE is supplied as an 80 mL fill in a 100 mL, single-use glass vial.
- Auxora 1.0 mg/kg (0.625 mL/kg): Medium dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
  CM-4620 Injectable Emulsion (CM4620-IE): Auxora is to be administered as an IV infusion and is supplied as a sterile, non-pyrogenic emulsion containing 1.6 mg/mL of the active pharmaceutical ingredient CM4620. CM4620-IE is supplied as an 80 mL fill in a 100 mL, single-use glass vial.
- Auxora 0.5 mg/kg (0.3125 mL/kg): Low dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
  CM-4620 Injectable Emulsion (CM4620-IE): Auxora is to be administered as an IV infusion and is supplied as a sterile, non-pyrogenic emulsion containing 1.6 mg/mL of the active pharmaceutical ingredient CM4620. CM4620-IE is supplied as an 80 mL fill in a 100 mL, single-use glass vial.
- Placebo (1.25, 0.625, or 0.3125 mL/kg): Patients randomized to placebo received one of three following volumes (1.25 mL/kg, 0.625 mL/kg, and 0.3125 mL/kg. Although patients are randomly assigned to the three volumes, all patients randomized to placebo are analyzed together as one arm. Placebo was administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Placebo: Matching Placebo is administered as an IV infusion and is supplied as a sterile, non-pyrogenic emulsion carrier containing no active pharmaceutical ingredient. Placebo is supplied as an 80 mL fill in a 100 mL single-use vial and contains the same ingredients as Auxora except that it does not contain CM4620.
Period: Overall Study
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Started | 54 | 56 | 53 | 53
Completed (* All 7 patients noted as "Lost to Follow-up" were known to be alive at Day 30 based on public records. * Of the 6 patients noted to have withdrawn consent prior to Day 30, 4 were known to be alive at Day 30 based on public records, 1 was known to have died based on public records, and 1 had unknown status (no public record).) | 49 | 53 | 51 | 49
Not Completed | 5 | 3 | 2 | 4
Not completed — Lost to Follow-up | 3 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 3
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two subjects were randomized but discharged before study drug could be administered. These two patients were excluded from all analysis.
Groups:
- Auxora 2.0 mg/kg (1.25 mL/kg): High dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
- Auxora 1.0 mg/kg (0.625 mL/kg): Medium dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
- Auxora 0.5 mg/kg (0.3125 mL/kg): Low dose Auxora, administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hour) for three consecutive days for a total of 3 doses.
- Placebo (1.25, 0.625, or 0.3125 mL/kg): Patients randomized to placebo received one of three following volumes (1.25 mL/kg, 0.625 mL/kg, and 0.3125 mL/kg. Although patients are randomly assigned to the three volumes, all patients randomized to placebo are analyzed together as one arm. Placebo was administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
- Total: Total of all reporting groups
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg) | Total
Number analyzed (Participants) | 53 | 56 | 52 | 53 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 40 | 47 | 179
  >=65 years | 5 | 12 | 12 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.58 (15.311) | 47.41 (16.876) | 49.23 (16.131) | 44.79 (15.181) | 46.26 (15.943)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 20 | 20 | 83
  Male | 33 | 33 | 32 | 33 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 14 | 13 | 45
  Not Hispanic or Latino | 42 | 46 | 38 | 39 | 165
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 16 | 17 | 16 | 20 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 13 | 10 | 8 | 8 | 39
  White | 21 | 26 | 22 | 15 | 84
  More than one race | 3 | 3 | 6 | 8 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 37 | 36 | 150
  India | 16 | 16 | 15 | 17 | 64
Etiology [Count of Participants; unit: Participants]
  Alcohol | 26 | 25 | 22 | 18 | 91
  Biliary | 8 | 11 | 10 | 14 | 43
  Drug Induced | 1 | 1 | 0 | 0 | 2
  Hypertriglyceridemia | 4 | 4 | 5 | 9 | 22
  Surgery/Trauma | 0 | 0 | 1 | 0 | 1
  Other | 4 | 4 | 4 | 4 | 16
  Unknown | 10 | 11 | 10 | 8 | 39
High Hematocrit (>/= 44 males; >/= 40 females) [Count of Participants; unit: Participants] | 23 | 25 | 24 | 20 | 92
Balthazar score D or E [Count of Participants; unit: Participants] — Balthazar score was based on screening CECT, as determined by central reading. Balthazar score grades the degree of pancreatitis, with A being best/normal and E being worst, as follows:
  A--normal pancreas, B--enlargement of pancreas, C--inflammatory changes in pancreas and peripancreatic fat, D--ill-defined single peripancreatic fluid collection, E--two or more poorly defined peripancreatic fluid collections
  Participants | 36 | 36 | 38 | 35 | 145
Abdominal Guarding or Rebound [Count of Participants; unit: Participants] | 38 | 44 | 35 | 37 | 154

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Solid Food Tolerance, With gMCP Modeling Analysis for Dose-response Relationship
Description: Time to Solid Food Tolerance (TSFT): Number of hours from date/time of SFISD to date/time patient receives a solid meal that is tolerated, defined as eating >/=50% of a low fat >/= 500-calorie solid meal w/o increase in abdominal pain or vomiting within 2 hours of mealtime.
  If patient was discharged w/o tolerating solid food, the daily record of the modified ANMS Gastrointestinal Cardinal Symptom Index Daily Diary (mGCSI-DD) at or after hospital discharge was used to calculate TSFT. For these patients, TSFT date/time was considered to be 8am on the first of 3 consecutive days where the following criteria were met in mGCSI-DD: no vomiting, no or mild nausea, no or mild inability to finish a normal sized meal, no or mild abdominal pain.
  gMCP-Mod: Generalized Multiple Comparisons and Modeling--3 steps: 1) Hazard ratio (dose vs placebo) using stratified Cox regression w/ stratification by sex and hematocrit (high/low). 2) Multiple contrast test. 3) Find best-fit dose-response model.
Time Frame: from start of first infusion of study drug (SFISD) through day 30
Population: Analysis for all treated patients and the high hematocrit subgroup are presented.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Hours
  All Patients | 67.0 [39.0 to 91.0] | 64.0 [43.0 to 93.0] | 78.0 [39.0 to 118.0] | 66.0 [44.0 to 116.0]
  High Hematocrit subgroup: number analyzed (Participants) | 23 | 25 | 24 | 20
  High Hematocrit subgroup | 67.0 [26.0 to 95.0] | 64.0 [20.0 to 101.0] | 78.0 [37.0 to 167.0] | 113.5 [40.0 to 187.0]
Statistical Analysis 1: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); The purpose of this analysis is to determine whether a dose-response relationship exists, with multiple possible models (Emax and sigEmax) being tested. gMCP-Mod analysis (Generalized Multiple Comparisons and Modeling) was performed in 3 steps as described in the SAP: 1) Hazard ratio (each dose vs placebo) using stratified Cox regression w/ stratification by sex and hematocrit (high/low HCT). 2) Multiple contrast test. 3) Find best-fit dose-response model. Emax model analysis is shown here; Test type: Other — The null hypothesis of flat dose-response relationship as compared to placebo for the primary efficacy endpoint was tested against the alternative hypothesis of a non-constant dose-response curve using a multiple contrast test as described in the gMCP-Mod methodology. The contrast test statistic is a linear combination of the optimal contrast coefficients corresponding to the dose-response curve model (Emax or sigEmax) with the hazard ratio obtained at each individual dose; p = 0.3184, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model based on all 3 dosage data points, not just the 0.5mg/kg point presented here; See Statistical Analysis 2 and 3 for the other two data points (1.0mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.0415
Statistical Analysis 2: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3184, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model based on all 3 dosage data points, not just the 1.0mg/kg point presented here; See Statistical Analysis 1 and 3 for the other two data points (0.5mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = .1225
Statistical Analysis 3: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3184, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model based on all 3 dosage data points, not just the 2.0mg/kg point presented here; See Statistical Analysis 1 and 2 for the other two data points (0.5mg/kg and 1.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.2080
Statistical Analysis 4: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); The purpose of this analysis is to determine whether a dose-response relationship exists, with multiple possible models (Emax and sigEmax) being tested. gMCP-Mod analysis (Generalized Multiple Comparisons and Modeling) was performed in 3 steps as described in the SAP: 1) Hazard ratio (each dose vs placebo) using stratified Cox regression w/ stratification by sex and hematocrit (high/low HCT). 2) Multiple contrast test. 3) Find best-fit dose-response model. sigEmax model analysis is shown here; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2265, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the sigEmax curve model based on data points for all 3 dosages, not just the 0.5mg/kg point presented here; See Statistical Analysis 5 and 6 for the other two data points (1.0mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.0415
Statistical Analysis 5: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2265, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the sigEmax curve model based on data points for all 3 dosages, not just the 1.0mg/kg point presented here; See Statistical Analysis 4 and 6 for the other two data points (0.5mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.1225
Statistical Analysis 6: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2265, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the sigEmax curve model based on data points for all 3 dosages, not just the 2.0mg/kg point presented here; See Statistical Analysis 4 and 5 for the other two data points (0.5mg/kg and 1.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.2080
Statistical Analysis 7: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); The purpose of this analysis is to determine whether a dose-response relationship exists for only the subset of patients with high HCT. Multiple possible models (Emax and sigEmax) were tested. gMCP-Mod (Generalized Multiple Comparisons & Modeling) analysis was performed in 3 steps as described in the SAP: 1) Hazard ratio (each dose vs placebo) using stratified Cox regression, stratification by sex 2) Multiple contrast test 3) Find best-fit dose-response model. Emax model analysis is shown here; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0764, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model for high HCT based on all 3 dosage data points, not just the 0.5mg/kg point shown here; See Statistical Analysis 8 and 9 for the other two data points (1.0mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.2671
Statistical Analysis 8: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 7]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0764, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model for high HCT based on all 3 dosage data points, not just the 1.0mg/kg point shown here; See Statistical Analysis 7 and 9 for the other two data points (0.5mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.6561
Statistical Analysis 9: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 7]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0764, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to the fit of the Emax curve model for high HCT based on all 3 dosage data points, not just the 2.0mg/kg point shown here; See Statistical Analysis 7 and 8 for the other two data points (0.5mg/kg and 1.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.4668
Statistical Analysis 10: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); The purpose of this analysis is to determine whether a dose-response relationship exists for the subset of patients with high HCT. Multiple possible models (Emax and sigEmax) were tested. gMCP-Mod (Generalized Multiple Comparisons & Modeling) analysis was performed in 3 steps as described in the SAP: 1) Hazard ratio (each dose vs placebo) using stratified Cox regression, stratification by sex 2) Multiple contrast test 3) Find best-fit dose-response model. sigEmax model analysis is shown here; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0574, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model for high HCT based on all 3 dosage data points, not just the 0.5mg/kg point shown here; See Statistical Analysis 11 and 12 for the other two data points (1.0mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.2671
Statistical Analysis 11: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 10]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0574, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model for high HCT based on all 3 dosage data points, not just the 1.0mg/kg point shown here; See Statistical Analysis 10 and 12 for the other two data points (0.5mg/kg and 2.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.6561
Statistical Analysis 12: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg) vs Placebo (1.25, 0.625, or 0.3125 mL/kg); [analysis description as in outcome 1, analysis 10]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0574, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model for high HCT based on all 3 dosage data points, not just the 2.0mg/kg point shown here; See Statistical Analysis 10 and 11 for the other two data points (0.5mg/kg and 1.0mg/kg) that are part of this same curve and p-value analysis; Hazard Ratio, log = 0.4668

2. Secondary Outcome: Percentage of Patients With New Onset Severe Respiratory Failure, With gMCP Modeling Analysis for Dose-response Relationship
Description: Analysis of patients without respiratory failure at the time of randomization (defined as a P/F ratio ≤300 measured by an arterial blood gas or imputed from pulse oximetry) who later developed severe respiratory failure during the course of the study.
Time Frame: from enrollment and through day 30
Population: Only the subset of patients without respiratory failure at the time of randomization (defined as a P/F ratio ≤300 measured by an arterial blood gas or imputed from pulse oximetry) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 50 | 52 | 48 | 47
Participants | 0 | 0 | 4 | 4
Statistical Analysis 1: Comparison: Placebo (1.25, 0.625, or 0.3125 mL/kg); Analysis to determine whether a dose-response relationship exists. Multiple possible models (Emax and sigEmax) were tested using gMCP-Mod (Generalized Multiple Comparisons & Modeling) analysis, performed in 3 steps as described in the SAP: 1) Odds ratio between each dose using logistic regression, with treatment, sex, and risk for organ failure (high/low HCT) as covariates 2) Multiple contrast test 3) Find best-fit dose-response model. Emax model analysis is shown here; Test type: Other — The null hypothesis of flat dose-response relationship as compared to placebo for the primary efficacy endpoint was tested against the alternative hypothesis of a non-constant dose-response curve using a multiple contrast test as described in the gMCP-Mod methodology. The contrast test statistic is a linear combination of the optimal contrast coefficients corresponding to the dose-response curve model (Emax or sigEmax) with the logit of rate of severe respiratory failure at each individual dose; p = 0.2379, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the Emax curve model based on all 4 dosage data points, not just the placebo data point shown here; See Statistical Analysis 2, 3, & 4 for the other data points (0.5mg/kg, 1.0mg/kg, and 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -2.3604
Statistical Analysis 2: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2379, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the Emax curve model based on all 4 dosage data points, not just the 0.5mg/kg data point shown here; See Statistical Analysis 1, 3, & 4 for the other data points (placebo, 1.0mg/kg, & 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -2.5078
Statistical Analysis 3: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2379, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the Emax curve model based on all 4 dosage data points, not just the 1.0mg/kg data point shown here; See Statistical Analysis 1, 2, & 4 for the other data points (placebo, 0.5mg/kg, & 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -4.8340
Statistical Analysis 4: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2379, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the Emax curve model based on all 4 dosage data points, not just the 2.0mg/kg data point shown here; See Statistical Analysis 1, 2, & 3 for the other data points (placebo, 0.5mg/kg, & 1.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -4.7657
Statistical Analysis 5: Comparison: Placebo (1.25, 0.625, or 0.3125 mL/kg); Analysis to determine whether a dose-response relationship exists. Multiple possible models (Emax and sigEmax) were tested using gMCP-Mod (Generalized Multiple Comparisons & Modeling) analysis, performed in 3 steps as described in the SAP: 1) Odds ratio between each dose using logistic regression, with treatment, sex, and risk for organ failure (high/low HCT) as covariates 2) Multiple contrast test 3) Find best-fit dose-response model. SigEmax model analysis is shown here; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0291, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model based on all 4 dosage data points, not just the placebo data point shown here; See Statistical Analysis 6, 7, & 8 for the other data points (0.5mg/kg, 1.0mg/kg, and 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -2.3604
Statistical Analysis 6: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg); [analysis description as in outcome 2, analysis 5]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0291, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model based on all 4 dosage data points, not just the 0.5mg/kg data point shown here; See Statistical Analysis 5, 7, & 8 for the other data points (placebo, 1.0mg/kg, & 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -2.5078
Statistical Analysis 7: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg); [analysis description as in outcome 2, analysis 5]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0291, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model based on all 4 dosage data points, not just the 1.0mg/kg data point shown here; See Statistical Analysis 5, 6, & 8 for the other data points (placebo, 0.5mg/kg, & 2.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -4.8340
Statistical Analysis 8: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0291, Mixed Models Analysis — p-value adjusted for multiple comparisons. Test is based on significance level of one-sided 15%.The p-value shown here relates to fit of the sigEmax curve model based on all 4 dosage data points, not just the 2.0mg/kg data point shown here; See Statistical Analysis 5, 6, & 7 for the other data points (placebo, 0.5mg/kg, & 1.0mg/kg) that are part of this same curve and p-value analysis; Odds Ratio, log = -4.7657

3. Secondary Outcome: Incidence, Severity, and Duration of Organ Failure
Description: The incidence, severity and duration of organ failure was defined by the development of severe respiratory failure or severe renal failure or severe cardiac failure. The proportion of patients who developed each type of organ failure, or multi-organ failure (more than 1 organ failure), was analyzed.
Time Frame: from enrollment and through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants
  Any severe organ failure | 2 | 2 | 5 | 5
  Severe respiratory failure | 2 | 2 | 5 | 4
  Severe renal failure | 0 | 1 | 2 | 1
  Severe cardiac failure | 1 | 1 | 3 | 1

4. Secondary Outcome: Solid Food Tolerance
Description: Number (and percentage) of patients who tolerated solid food at 48hrs, 72hrs, and 96hrs from start of first infusion of study drug, as well as at time of first discharge from hospital
Time Frame: from SFISD to 48 hours, 72 hours and 96 hours and at time of hospital discharge (up to 30 days after SFISD)
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants
  48hrs | 23 | 26 | 23 | 21
  72hrs | 27 | 30 | 25 | 30
  96hrs | 37 | 35 | 31 | 30
  Hospital Discharge | 44 | 41 | 39 | 42

5. Secondary Outcome: Time to Medically Indicated Discharge
Description: The time (in hours) to medically indicated discharge, defined as the number of days from the SFISD to the first date of meeting the criteria below:
  * the patient tolerated solid food, as defined by the main analytical approach; and
  * abdominal pain was controlled or resolved, which was defined by a reduction in pain, as assessed by the PNRS scale, of ≥50% from the peak level in the first 24 hours and no use of opioids; and
  * no clinical evidence of an infection requiring continued hospitalization. Kaplan-Meier (K-M) estimates of median time to medically indicated discharge are shown.
Time Frame: from start of first infusion of study drug through time of hospital discharge or through Day 30, whichever occurs first
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
hours | 89 [48 to 118] | 104.5 [73 to 164] | 109.5 [82 to 164] | 104 [67 to 144]

6. Secondary Outcome: Length of Stay in the Hospital
Description: Number of days in the hospital during the first 30 Days of the Study from the SFISD (start of first infusion of study drug) while still alive, for any reason. Includes ICU stay and readmissions. The number of days in the hospital before the patient's death was used in the analysis.(Note: there was only 1 patient death in this study, in the 1.0 mg/kg Auxora group)
Time Frame: from admission date into the hospital until discharge date from the hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
days | 5.9 (3.77) | 5.9 (4.46) | 7.6 (6.54) | 7.1 (5.87)

7. Secondary Outcome: Re-hospitalization for Acute Pancreatitis by Day 30
Description: The proportion of patients who were re-hospitalized for either acute pancreatitis, or the development of pancreatic necrosis/necrotizing pancreatitis through the Day 30 visit.
Time Frame: time from initial date of hospital discharge through date of re-hospitalization through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants
  All rehospitalizations due to AP | 4 | 3 | 1 | 0
  Cause of AP rehospitalization - alcohol | 2 | 2 | 0 | 0
  Cause of AP rehospitalization - biliary | 1 | 0 | 1 | 0
  Cause of AP rehospitalization - abdominal pain (from AP) | 1 | 0 | 0 | 0
  Cause of AP rehospitalization - hypertriglyceridemia | 0 | 1 | 0 | 0

8. Secondary Outcome: Change in Severity of Acute Pancreatitis by CTSI Score From Screening to Day 30
Description: Independent reviewers performed a blinded central review of Contrast Enhanced Computed Tomography (CECT) imaging data, or MRI imaging data, obtained at the Screening and Day 30 visits to assess the Computed Tomography Severity Index (CTSI). Review was performed by two independent radiologists (primary review) using a consensus methodology. The CTSI scoring uses a combination of Balthazar score grading of pancreatitis (A-E) and grading the extent of pancreatic necrosis (none, ≤30%, >30-50%, or >50%) to designate AP as mild, moderate, or severe.
  Proportion of patients with moderate or severe AP by CTSI score at baseline who became mild AP at Day 30, and the proportion of patients with mild AP by CTSI at baseline who had moderate or severe AP at Day 30 were analyzed.
Time Frame: From informed consent through day 30
Population: Patients were divided into two subgroups for this analysis: those with Moderate or Severe AP by CTSI score at baseline, and those with Mild AP by CTSI score at baseline. Analysis only includes subjects with non-missing Screening and Day 30 Visit (or post-treatment unscheduled visit) CTCE reading results.
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 38 | 49 | 45 | 41
Participants
  Patients with Moderate or Severe AP at baseline who had Mild AP at Day 30 (by CTSI score): number analyzed (Participants) | 23 | 26 | 24 | 25
  Patients with Moderate or Severe AP at baseline who had Mild AP at Day 30 (by CTSI score) | 10 | 8 | 12 | 14
  Patients with Mild AP at baseline who had Moderate or Severe AP at Day 30 (by CTSI score): number analyzed (Participants) | 15 | 23 | 21 | 16
  Patients with Mild AP at baseline who had Moderate or Severe AP at Day 30 (by CTSI score) | 0 | 2 | 2 | 0

9. Secondary Outcome: Development of Pancreatic Necrosis ≥30% and >50%
Description: Development of pancreatic necrosis ≥30% and >50% in patients who had no pancreatic necrosis at screening (Note: There were no patients with pancreatic necrosis at screening in any of the treatment groups.)
Time Frame: from enrollment CECT through Day 30 CECT
Population: Only subjects with non-missing Screening and Day 30 Visit (or post-treatment unscheduled visit) CTCE reading results were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 39 | 49 | 45 | 41
Participants
  Pancreatic Necrosis >50% | 1 | 1 | 1 | 0
  Pancreatic Necrosis 30% to 50% | 0 | 0 | 1 | 0

10. Secondary Outcome: The Persistence of SIRS ≥48 Hours After the SFISD
Description: The proportion of patients who developed persistence of SIRS ≥48 Hours after the SFISD analyzed through Day 30. If the patient was discharged before 48 Hours after the SFISD, the last available post-treatment data was used to define the SIRS status at 48 hours after the SFISD based on the LOCF method.
Time Frame: from SFISD through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants | 11 | 8 | 15 | 13

11. Secondary Outcome: Mortality by Day 30
Description: Mortality was assessed from randomization through Day 30
Time Frame: from randomization and through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants | 0 | 1 | 0 | 0

12. Secondary Outcome: Change in Pain Score
Description: Mean change in Pain Numeric Rating Score (PNRS) from baseline (time of screening). In patients who were able to self-report their pain, the PNRS was used to grade the severity of the abdominal pain. Patients were asked, "On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable, how would you rate your pain RIGHT NOW." It was also recorded if an opioid analgesic had been given in the 2 hours prior to the PNRS determination.
Time Frame: from enrollment through day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
score on a scale
  Change from Baseline at 48hrs | -3.3 (3.33) | -3.2 (2.98) | -3.2 (3.22) | -3.1 (3.10)
  Change from Baseline at 72hrs | -4.1 (3.49) | -3.8 (3.18) | -3.8 (3.71) | -3.7 (3.18)
  Change from Baseline at 96hrs | -4.6 (3.26) | -4.5 (3.87) | -3.1 (3.21) | -3.6 (2.29)

13. Other Pre Specified Outcome: Win Ratio for Auxora vs. Placebo
Description: The win ratio compares effectiveness of each Auxora dose group with the placebo group. It is calculated by dividing the total number of wins by the total number of losses, with a win ratio >1 indicating better outcomes for Auxora treatment. Comparison between placebo and Auxora outcomes was performed in a hierarchical manner, in the following order: 1. Mortality (see Outcome Measure 11), 2. New Onset Severe Respiratory Failure (see Outcome Measure 2), 3. New Onset Necrotizing Pancreatitis at Day 30 (see Outcome Measure 18), and 4. Time to Medically Indicated Discharge (see Outcome Measure 5).
  Stratification was performed by sex (male or female) and then by HCT (higher or lower).
  Subjects with respiratory failure at baseline were imputed as a non-event. Subjects with missing necrotizing pancreatitis evaluation or positive necrotizing pancreatitis at screening were imputed as a non-event. Subjects missing a necrotizing pancreatitis evaluation at Day 30 were imputed as a non-event.
Time Frame: from randomization through Day 30
Measure: Number (95% Confidence Interval); unit: Win Ratio
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52
Win Ratio
  Stratified Win Ratio - ALL | 1.640 [1.030 to 2.612] | 1.177 [0.740 to 1.871] | 1.123 [0.708 to 1.781]
  Stratified Win Ratio - High HCT | 1.507 [0.741 to 3.063] | 1.241 [0.586 to 2.627] | 1.200 [0.596 to 2.415]
  Stratified Win Ratio - Balthazar D or E | 2.071 [1.135 to 3.779] | 1.501 [0.827 to 2.724] | 1.613 [0.922 to 2.824]
Statistical Analysis 1: Comparison: Auxora 2.0 mg/kg (1.25 mL/kg); Test type: Superiority; p = 0.0372, Finkelstein-Schoenfeld
Statistical Analysis 2: Comparison: Auxora 1.0 mg/kg (0.625 mL/kg); Test type: Superiority; p = 0.4918, Finkelstein-Schoenfeld
Statistical Analysis 3: Comparison: Auxora 0.5 mg/kg (0.3125 mL/kg); Test type: Superiority; p = 0.6224, Finkelstein-Schoenfeld

14. Other Pre Specified Outcome: Development of Infected Pancreatic Necrosis
Description: Exploratory. Percentage of Patients with Infected Pancreatic Necrosis at Day 30 after SFISD.
Time Frame: from end of first infusion of study drug through Day 30 CECT
Population: Count and percentage is based on the number of subjects with non-missing Screening and Day 30 Visit (or post-treatment unscheduled visit) CTCE reading results.
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 39 | 49 | 45 | 41
Participants | 1 | 0 | 0 | 1

15. Other Pre Specified Outcome: Development of Sepsis
Description: Exploratory. Count of patients who experienced sepsis after SFISD.
Time Frame: from end of first infusion of study drug through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 53 | 56 | 52 | 53
Participants | 0 | 2 | 3 | 1

16. Other Pre Specified Outcome: Change in ANC/ALC Ratio and IL-6 Levels
Description: Exploratory analysis of serum biomarkers.
Time Frame: from randomization through day 30
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Urine NGAL
Description: Exploratory analysis of urine biomarker NGAL
Time Frame: from randomization through day 30
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Number of Patients That Developed Any New Onset Necrotizing Pancreatitis by Day 30
Description: The number of patients who had no necrotizing pancreatitis at screening, and developed any amount of necrotizing pancreatitis based on the Day 30 visit CECT reading results.
Time Frame: From SFISD to Day 30
Population: Analysis includes only patients who had a CECT at screening that showed no necrotizing pancreatitis, and who also had a non-missing Day 30 visit (or post-treatment unscheduled visit) CECT
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
Number analyzed (Participants) | 37 | 49 | 44 | 46
Participants | 11 | 27 | 24 | 17

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events daily, from randomization to their final visit. Documentation of each patient's adverse events continued until the patient died, the patient withdrew consent, or the patient's participation in the study ended. For patients who completed the study, the last AE assessment performed on Day 30 visit, which was scheduled 30 days after start of first infusion of study drug +/- 5 days.
Groups:
- Placebo (1.25, 0.625, or 0.3125 mL/kg): Patients randomized to placebo received one of three following volumes (1.25 mL/kg, 0.625 mL/kg, and 0.3125 mL/kg. Although patients are randomly assigned to the three volumes, all patients randomized to placebo are analyzed together as one arm. Placebo was administered intravenously over 4 hours at a constant rate of infusion. Infusions were administered every 24 hours (±1 hours) for three consecutive days for a total of 3 doses.
  Placebo: Matching Placebo is administered as an IV infusion and is supplied as a sterile, non-pyrogenic emulsion carrier containing no active pharmaceutical ingredient. Placebo is supplied as an 80 mL fill in a 100 mL single-use vial. Placebo contains the same ingredients as Auxora except that it does not contain CM4620.
Arm/Group | Auxora 2.0 mg/kg (1.25 mL/kg) | Auxora 1.0 mg/kg (0.625 mL/kg) | Auxora 0.5 mg/kg (0.3125 mL/kg) | Placebo (1.25, 0.625, or 0.3125 mL/kg)
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/56 | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 8/53 | 12/56 | 13/52 | 6/53
Other Adverse Events (participants affected / at risk) | 22/53 | 32/56 | 26/52 | 23/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auxora 2.0 mg/kg (1.25 mL/kg) (N=53) | Auxora 1.0 mg/kg (0.625 mL/kg) (N=56) | Auxora 0.5 mg/kg (0.3125 mL/kg) (N=52) | Placebo (1.25, 0.625, or 0.3125 mL/kg) (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (3) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripancreatic fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endoscopic ultrasound (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auxora 2.0 mg/kg (1.25 mL/kg) (N=53) | Auxora 1.0 mg/kg (0.625 mL/kg) (N=56) | Auxora 0.5 mg/kg (0.3125 mL/kg) (N=52) | Placebo (1.25, 0.625, or 0.3125 mL/kg) (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6) | 3 (3) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (4) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripancreatic fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesenteric cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudocyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Murphy's sign positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall submit copies of the proposed results communications to the Sponsor at least 30 days in advance of the submission of any proposed publication to a journal, editor, or other third party. Sponsor may request that Confidential Information (other than Study Data) be removed from communications, or that the PI refrain from publication for an additional 60 days in order for patent application(s) directed to the patentable subject matter to be filed with the appropriate patent office(s).

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04681066/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04681066/SAP_001.pdf